CLINICAL TRIAL: NCT05150262
Title: Urinary Procedures Performed by Gynecologists, Results and Learning Curves.
Acronym: URINA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8417
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Gynecologic Cancer; Endometriosis
Keywords: Gynecologic Cancer; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary procedures such as placing a JJ catheter, performing a psoic bladder, a Bricker technique or even a partial cystectomy are relatively frequent procedures in the context of the surgical management of gynecological cancer or endometriosis in order to obtain maximum reduction in oncology, or to overcome all endometriotic lesions when they affect the urinary tract. However, gynecological surgeons are not always trained in these specific procedures, the learning of which is crucial in the optimal management of these patients.

The aim of the research is to describe the surgical experience in terms of urinary actions (JJ catheter placement, psoic bladder, Bricker technique, cystectomy) over the past 10 years and determine a learning curve for a surgical team made up of only gynecological surgeons

ELIGIBILITY:
Inclusion criteria:

* Adult woman (≥18 years old)
* Woman with gynecological cancer or endometriosis, having undergone surgery between 01/01/2010 and 04/30/2021 at Strasbourg University Hospital
* With the performance of urological procedures during the operation performed by a surgical team composed of a gynecological surgeon
* Woman who did not express her opposition to the reuse of her data for the purposes of this research.

Exclusion criteria:

* Woman who expressed her opposition to participating in the study
* Surgery performed by a team of surgeons not composed exclusively of gynecologists

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult woman with gynecological cancer or endometriosis, having undergone surgery between 01/01/2010 and 04/30/2021 at Strasbourg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Describe the surgical experience in terms of urinary procedures (JJ catheter placement, psoic bladder, Bricker's technique, cystectomy) over the past 10 years | Files analysed retrospectively from January 01, 2010 to April 30, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Lise LECOINTRE, MD, Principal Investigator — Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France